CLINICAL TRIAL: NCT00361712
Title: Effect of Preemptive Epidural Analgesia in Labor on Pro and Anti-inflammatory Cytokine Production in a Mother and a Newborn
Brief Title: Effect of Preemptive Epidural Analgesia in Labor on Cytokine Production
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, sharonorbach, Dr, Rabin Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 003692
Record Dates: First submitted 2006-08-06; First posted 2006-08-08 (Estimated); Results first posted 2018-03-12 (Actual); Last update posted 2018-04-09 (Actual); Status verified 2018-03

CONDITIONS: Obstetric Pain
Keywords: Epidural; analgesia; labor; cytokines
MeSH Terms: conditions — Labor Pain; Agnosia | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Preemptive epidural analgesia (Experimental): Parturients will receive epidural analgesia immediately upon arrival in the labor ward before onset of painful contractions (VAS<3).
  Interventions: Procedure: Preemptive epidural analgesia
- Standard of care (Active Comparator): Parturients with cervical dilatation and painful labor (VAS >5) will receive epidural analgesia as soon as possible
  Interventions: Drug: Standard of care

INTERVENTIONS:
Procedure: Preemptive epidural analgesia — Parturients will receive early epidural analgesia before onset of painful contractions as oppose to standard of care in which parturients receive epidural analgesia with onset of painful contractions.
  Arms: Preemptive epidural analgesia
Drug: Standard of care — Epidural analgesia with parturients with cervical dilatation and painful labor (VAS >5)
  Arms: Standard of care

SUMMARY:
During labor there is an increased production of inflammatory mediators called cytokines. Higher concentration of certain cytokines has been linked to adverse neonatal and maternal outcomes.

Epidural analgesia is commonly performed after the parturient feels labor pain.

We hypothesis that preemptive epidural analgesia (initiated before labor pain begins)can influence the production of cytokines.

DETAILED DESCRIPTION:
The interrelationship between vaginal labor, cytokine production, and epidural analgesia is unknown. Vaginal delivery is thought to induce a maternal inflammatory response. Though epidural analgesia during labor was found to significantly influence peripartum maternal and newborn interleukin concentrations, these studies did not address at what stage epidural analgesia was performed. Preemptive analgesia has been found to be associated with attenuated proinflammatory cytokines, at least in the postoperative period.

Healthy ASA I term parturients (>37 weeks) being accepted into delivery ward and wanting epidural analgesia will be studied.

Parturients will be divided into two groups:

* Group I- those who have painless contractions awaiting augmentation of labor.
* Group II- parturients with cervical dilatation and painful labor (VAS >5).

Parturients in Group I will be given epidural analgesia immediately upon arrival in the labor ward before onset of painful contractions (VAS<3). Parturients in Group 2 will be given epidural analgesia as soon as possible.

Epidural analgesia protocol will be identical for both groups: graduated doses of bupivicaine 0.1% 15cc and 100 mcg fentanyl followed by patient controlled analgesia at a concentration of bupivicaine 0.1% and fentanyl 2 mcg/cc delivered at 10cc per hour with possible boluses of 5 cc every ten minutes.

Maternal serum will be drawn before epidural insertion and 18-24 hours after delivery. Placental blood will be drawn after delivery.

These blood sample will be assessed for IL-1Beta, TNF alpha, IL-1ra, IL-2, Il-6, IL-8, IL-10, IL-18.

The patient's chart will be prospectively analyzed for demographic information about parturient and complications and progress of labor.

ELIGIBILITY:
Inclusion Criteria:

1. Age>18
2. Singleton pregnancy with no known fetal malformations
3. Above or equal to 38 weeks of pregnancy

Exclusion Criteria:

1. Systemic medical illnesses
2. Chronic medications except for iron and vitamins
3. Women developing fever > 380C
4. Women with history of delivery of children with cerebral palsy
5. History of infertility
6. Premature contractions

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2006-07; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Orbach-Zinger, M.D., Study Director — Department of Anesthesiology, Rabin Medical Center/Beilinson Hospital
Locations (1):
- Rabin Medical Center/Beilinson Campus, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Women in labor were recruited for the study at entry to the triage area of the delivery room of a major tertiary medical center from January to May 2006.
Groups:
- Randomized to Early Epidural Analgesia: Parturients were allocated to receive epidural analgesia immediately on admission, before the onset of painful contractions
- Randomized to Epidural Analgesia Upon Request: Parturient's pain was monitored every 15 min until it reached a level of >50 on the VAS and then epidural analgesia was initiated.
Period: Overall Study
Arm/Group | Randomized to Early Epidural Analgesia | Randomized to Epidural Analgesia Upon Request
Started | 20 | 21
Completed | 20 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Randomized to Early Epidural Analgesia | Randomized to Epidural Analgesia Upon Request | Total
Number analyzed (Participants) | 20 | 21 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.5 (3.6) | 29.1 (4.9) | 30.5 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 21 | 41
  Male | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Israel | 20 | 21 | 41

OUTCOME MEASURES:

1. Primary Outcome: Maternal Cytokine IL-10 Levels of pg/ml Upon Enrollment
Description: Maternal serum cytokine IL-10 levels of pg/ml measured upon enrollment
Time Frame: Right after enrollment
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Randomized to Early Epidural Analgesia | Randomized to Epidural Analgesia Upon Request
Number analyzed (Participants) | 20 | 21
pg/ml | 12.7 (4.5) | 14.2 (7)

2. Primary Outcome: Maternal Cytokine of pg/ml IL-10 Levels 24 Hours After Delivery
Description: Maternal serum cytokine levels of pg/ml IL-10 as measured 24 hours after delivery
Time Frame: 24 hours after delivery
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Randomized to Early Epidural Analgesia | Randomized to Epidural Analgesia Upon Request
Number analyzed (Participants) | 20 | 21
pg/ml | 15.22 (5.6) | 16.77 (0)

3. Primary Outcome: Umbilical Cord Cytokine of pg/ml IL-10 Levels at Birth
Description: Umbilical cord cytokine IL-10 levels pg/ml as measured at delivery
Time Frame: At birth of parturients
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Randomized to Early Epidural Analgesia | Randomized to Epidural Analgesia Upon Request
Number analyzed (Participants) | 20 | 21
pg/ml | 1 (0.6) | 1.5 (1.3)

ADVERSE EVENTS:
Time Frame: Adverse events were recorded throughout study participation period four months
Arm/Group | Randomized to Early Epidural Analgesia | Randomized to Epidural Analgesia Upon Request
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/21
Other Adverse Events (participants affected / at risk) | 9/20 | 0/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Randomized to Early Epidural Analgesia (N=20) | Randomized to Epidural Analgesia Upon Request (N=21)
Hyoptension (Pregnancy, puerperium and perinatal conditions) | 4 | 0
meconium in the amniotic ﬂuid (Pregnancy, puerperium and perinatal conditions) | 5 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No